CLINICAL TRIAL: NCT02347189
Title: Melody(TM) Transcatheter Pulmonary Valve PB1016 Surveillance Study Implantation of the Medtronic Melody Transcatheter Pulmonary Valve PB1016 Using the Ensemble(TM) Transcatheter Delivery System in Patients With Dysfunctional RVOT Conduits
Brief Title: Melody PB1016 Surveillance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Heart Valves (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10154745DOC
Record Dates: First submitted 2014-09-12; First posted 2015-01-27 (Estimated); Results first posted 2017-11-29 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-10

CONDITIONS: Dysfunctional RVOT Conduits in Patients With Congenital Heart Defects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Melody TPV PB1016 (Other)
  Interventions: Device: Melody Transcatheter Pulmonary Valve PB1016

INTERVENTIONS:
Device: Melody Transcatheter Pulmonary Valve PB1016

SUMMARY:
Non-randomized, multi-center, prospective surveillance study to investigate and assess the residual risks, and to confirm the currently established safety and performance of the Melody TPV PB1016.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible to receive Melody TPV PB1016 per current Instructions for Use (IFU) indications at time of study enrollment
* Patient (or patient's legally authorized representative) is willing to consent to participate in the study and will commit to completion of all follow-up requirements.

Exclusion Criteria:

* Implantation in the aortic, tricuspid, or mitral position
* Venous anatomy unable to accommodate a 22-Fr size introducer sheath
* Obstruction of the central veins
* Clinical or biological signs of infection including active endocarditis
* History of intravenous substance abuse
* Currently participating in an investigational drug or device study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2018-08-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (5):
  - University of California - Los Angeles, Los Angeles, California
  - Children's Hospital of Michigan, Detroit, Michigan
  - Nationwide Childrens Hospital, Columbus, Ohio
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Childrens and Regional Hospital, Seattle, Washington
- Landes-Kinderklinik, Linz, Austria
- Stollery Childrens Hospital, Edmonton, Alberta, Canada
- Hospital General Universitario Gregorio Marañón, Madrid, Spain

REFERENCES:
- [Derived] Morray BH, Jones TK, Coe JY, Gitter R, Martinez JZ, Turner DR, Gray RG, Lung TH, Berman DP, Levi DS. Implantation of the Melody transcatheter pulmonary valve PB1016 in patients with dysfunctional right ventricular outflow tract conduits. Catheter Cardiovasc Interv. 2019 Feb 15;93(3):474-480. doi: 10.1002/ccd.27974. Epub 2018 Nov 12. PMID 30419603

RESULTS

PARTICIPANT FLOW:
Groups:
- Melody PB1016 Subjects Consented (i.e. Enrolled): This study is comprised of a single arm of subjects consented (i.e. enrolled) into the trial. All enrolled subjects were intended to be treated with the Melody TPV PB1016 device. Not all subjects enrolled ultimately received the device.
Period: Overall Study
Arm/Group | Melody PB1016 Subjects Consented (i.e. Enrolled)
Started (Number of subjects consented) | 39
Catheterized (Number of subject catheterized with the intent of implant Melody TPV PB1016) | 39
Implanted (Number of subjects implanted with a Melody TPV PB1016) | 30
Implanted > 24 Hours (Number of subjects implanted successfully for at least 24 hours) | 30
Completed (Number of subjects with evaluable data at 6 months) | 28
Not Completed | 11
Not completed — No implant attempted of study device | 9
Not completed — No primary outcome data available | 2

BASELINE CHARACTERISTICS:
Population: All subjects consented
Arm/Group | Melody PB1016 Subjects Consented (i.e. Enrolled)
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.2 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 25
Region of Enrollment [Number; unit: participants]
  Canada | 3
  Austria | 4
  United States | 29
  Spain | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Acceptable TPV Hemodynamic Function At 6 Months
Description: Acceptable TPV hemodynamic function at six months after successful TPV implantation which is determined as a composite of the following:
  * Mean Right Ventricular Outflow Tract (RVOT) gradient is less than or equal to 30 mmHg as measured by Continuous-wave Doppler (CW Doppler) echocardiography, and
  * Severity of pulmonary regurgitation less than moderate by CW Doppler echocardiography, and
  * Free from RVOT conduit reoperation or catheter re-intervention on the TPV at six months post-TPV implantation
Time Frame: 6 Months
Population: 28 subjects successfully implanted for greater than 24 hours (out of 30 total) had evaluable data at 6 months.
Measure: Count of Participants; unit: Participants
Groups:
- Implanted > 24 Hours Cohort: Subjects included in this analysis were those who were successfully implanted with a Melody TPV PB1016 for greater than 24 hours and had evaluable data at 6 months.
Arm/Group | Implanted > 24 Hours Cohort
Number analyzed (Participants) | 28
Participants | 25

2. Secondary Outcome: Number of Subjects With Acceptable TPV Hemodynamic Function At 1 Year
Description: Acceptable TPV hemodynamic function at 1 year after successful TPV implantation which is determined as a composite of the following:
  * Mean RVOT gradient is ≤ 30 mmHg as measured by CW Doppler
  * Severity of pulmonary regurgitation is less than moderate by Doppler echocardiography
  * Free from RVOT conduit reoperation or catheter re-intervention on the TPV at 1 year post-TPV implantation.
Time Frame: 1 Year
Population: 25 subjects successfully implanted for greater than 24 hours (out of 30 total) had evaluable data at 1 year.
Measure: Count of Participants; unit: Participants
Groups:
- Implanted > 24 Hours Cohort: Subjects included in this analysis were those who were successfully implanted with a Melody TPV PB1016 for greater than 24 hours and had evaluable data at 1 year.
Arm/Group | Implanted > 24 Hours Cohort
Number analyzed (Participants) | 25
Participants | 23

3. Secondary Outcome: Number of Subjects With Acceptable TPV Hemodynamic Function at 2 Years
Description: Acceptable TPV hemodynamic function at 2 years after successful TPV implantation which is determined as a composite of the following:
  * Mean RVOT gradient is ≤ 30 mmHg as measured by CW Doppler
  * Severity of pulmonary regurgitation is less than moderate by Doppler echocardiography
  * Free from RVOT conduit reoperation or catheter re-intervention on the TPV at 2 years post-TPV implantation.
Time Frame: 2 Years
Population: 27 subjects successfully implanted for greater than 24 hours (out of 30 total) had evaluable data at 2 years.
Measure: Count of Participants; unit: Participants
Groups:
- Implanted > 24 Hours Cohort: Subjects included in this analysis were those who were successfully implanted with a Melody TPV PB1016 for greater than 24 hours and had evaluable data at 2 years.
Arm/Group | Implanted > 24 Hours Cohort
Number analyzed (Participants) | 27
Participants | 25

4. Secondary Outcome: Number of Subjects With Serious Procedure-related and Device-related Adverse Events
Description: * Serious procedure-related adverse events at 1year and 2 years post-implant
  * Serious device-related adverse events at 1 year and 2 years post-implant
Time Frame: 1 Year, 2 Years
Measure: Count of Participants; unit: Participants
Groups:
- Catheterized Cohort: Procedure-related SAEs at 1 yr; Catheterized Cohort: Procedure-related SAEs at 2 Yrs: Subjects included in this analysis were those who went to the catheterization lab for implantation of a Melody PB1016.
- Implanted > 24 Hours Cohort: Device-related SAEs at 1 yr; Implanted > 24 Hours Cohort: Device-related SAEs at 2 Yrs: Subjects included in this analysis were those who were implanted with the Melody PB1016 > 24 hours.
Arm/Group | Catheterized Cohort: Procedure-related SAEs at 1 yr | Catheterized Cohort: Procedure-related SAEs at 2 Yrs | Implanted > 24 Hours Cohort: Device-related SAEs at 1 yr | Implanted > 24 Hours Cohort: Device-related SAEs at 2 Yrs
Number analyzed (Participants) | 39 | 39 | 30 | 30
Participants | 8 | 8 | 1 | 3

5. Secondary Outcome: Number of Subjects With Procedural Success
Description: A successful implant is defined as follows:
  * Melody TPV PB1016 is fixated within the desired location
  * RV-PA peak-to-peak gradient measured in the catheterization lab after Melody TPV PB1016 implantation is < 35 mmHg
  * No more than trace/trivial pulmonary regurgitation by angiography
  * Subject is free from explantation of the Melody TPV PB1016 at 24 hours post-implant.
Time Frame: At Time Of Procedure
Population: In one subject, the right ventricle to pulmonary artery (RV-PA) peak-to-peak gradient was not collected, leaving the overall number of evaluable subjects analyzed at 29 versus 30.
Measure: Count of Participants; unit: Participants
Groups:
- Implanted > 24 Hours Cohort: Subjects included in this analysis were those who were successfully implanted
Arm/Group | Implanted > 24 Hours Cohort
Number analyzed (Participants) | 29
Participants | 25

6. Secondary Outcome: Percentage of Participants Who Met Various Safety Parameters of the Melody TPV PB1016
Description: * Kaplan-Meier: Freedom from Stent Fracture
  * Kaplan-Meier: Freedom from re-intervention on the Melody TPV PB1016
  * Kaplan-Meier: Freedom from RVOT Conduit Operation
  * Kaplan-Meier: Freedom from Death (All-Cause)
Time Frame: 2 years
Measure: Number; unit: percentage of subjects
Groups:
- Implanted > 24 Hours Cohort / Freedom From Stent Fracture; Implanted > 24 Hours Cohort / Freedom From TPV Re-intervention; Implanted > 24 Hours Cohort / Freedom From All-Cause Mortality; Implanted > 24 Hours Cohort / Freedom From RVOT Reoperation: Subjects included in this analysis were those successfully implanted with a Melody TPV PB1016 for > 24 hours.
Arm/Group | Implanted > 24 Hours Cohort / Freedom From Stent Fracture | Implanted > 24 Hours Cohort / Freedom From TPV Re-intervention | Implanted > 24 Hours Cohort / Freedom From All-Cause Mortality | Implanted > 24 Hours Cohort / Freedom From RVOT Reoperation
Number analyzed (Participants) | 28 | 30 | 30 | 30
percentage of subjects | 96.4 | 96.7 | 100 | 96.7

ADVERSE EVENTS:
Time Frame: Adverse Event data are collected from the point of enrollment (consent signed) through a subject's 2 year visit.
Description: Serious Adverse Event:
  1. led to death,
  2. led to a serious deterioration in the health of the subject, resulting in
     1. a life-threatening illness or injury or
     2. a permanent impairment of a body structure or a body function or
     3. in-patient or prolonged hospitalization or
     4. medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function
  3. led to foetal distress, death or congenital abnormality/birth defect.
Arm/Group | Melody PB1016 Subjects Consented (i.e. Enrolled)
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 14/39
Other Adverse Events (participants affected / at risk) | 16/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melody PB1016 Subjects Consented (i.e. Enrolled) (N=39)
Atrial Flutter (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Cardiac Disorder (Cardiac disorders) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 1 (2)
Junctional Rhythm (Cardiac disorders) | 1 (1)
Pulmonary Valve Stenosis (Cardiac disorders) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Device Complication (General disorders) | 1 (1)
Device Rupture (General disorders) | 3 (3)
Endocarditis (Infections and infestations) | 3 (3)
Prosthetic Valve Endocarditis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Procedural Hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Central Nervous System Disorder* (Nervous system disorders) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melody PB1016 Subjects Consented (i.e. Enrolled) (N=39)
Congestive Heart Failure (Cardiac disorders) | 2 (2)
Tricuspid Regurgitation (Cardiac disorders) | 3 (3)
Gastrointestinal Disorder (Gastrointestinal disorders) | 3 (5)
Vomiting (Gastrointestinal disorders) | 2 (2)
Adverse Event (General disorders) | 7 (9)
Chest Pain (General disorders) | 3 (3)
Upper Repiratory Tract Infection (Infections and infestations) | 2 (2)
Vascular Access Complication (Injury, poisoning and procedural complications) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less